CLINICAL TRIAL: NCT03207737
Title: A Blended Residential/Telehealth Lifestyle Intervention to Improve Cardiovascular Health and Manage Pain in Adults With Spinal Cord Injury.
Brief Title: Mindfulness, Exercise and Nutrition To Optimize Resilience for Individuals With a Spinal Cord Injury.
Acronym: MENTOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Lakeshore Foundation (Other); The Craig H. Neilsen Foundation (Other)
Responsible Party: Principal Investigator, James Rimmer, Principal Investigator, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB-170123001
Record Dates: First submitted 2017-06-28; First posted 2017-07-05 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Spinal Cord Injuries
Keywords: Spinal Cord Injuries; SCI; Telehealth; Mindfulness; Nutrition; Exercise
MeSH Terms: conditions — Spinal Cord Injuries; Motor Activity | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MENTOR + Telehealth (Experimental): This group will complete baseline testing, the MENTOR (Mindfulness, Exercise, and Nutrition To Optimize Resilience) program, and 5-days post baseline testing before beginning a one-year telehealth program.
  Interventions: Behavioral: MENTOR + Telehealth
- Telehealth Only (Active Comparator): This group will complete baseline and 5-days post baseline testing before beginning a one-year telehealth program.
  Interventions: Behavioral: Telehealth Only

INTERVENTIONS:
Behavioral: MENTOR + Telehealth — Participants will live on campus for one week and complete the MENTOR program, which is a course about resilience and how nutrition, exercise and mindfulness help with resilience for individuals with a spinal cord injury. Different experts will cover the three main topics with lectures and application of knowledge through related activities. Participants will then begin a one-year telehealth program at home. The telehealth program will consist of readily available information focusing on nutrition, exercise and mindfulness for individuals with a spinal cord injury and a telehealth coach who will interact on the phone with the participants once every two weeks. This will continue for a total of 26 phone calls until the participant returns for 1-year follow-up testing.
  Arms: MENTOR + Telehealth
Behavioral: Telehealth Only — Participants will complete a one-year telehealth program at home. The telehealth program will consist of readily available information focusing on nutrition, exercise and mindfulness for individuals with a spinal cord injury and a telehealth coach who will interact on the phone with the participants once every two weeks. This will continue for a total of 26 phone calls until the participant returns for 1-year follow-up testing.
  Arms: Telehealth Only

SUMMARY:
The purpose of this study is to examine the effects of onsite and telehealth programs for individuals with spinal cord injury. The primary aim of this study is to compare the effectiveness of a blended 5-day onsite health promotion program followed by a 12-month telehealth package composed of exercise, nutrition, and mindfulness, to a 12-month telehealth-only package in individuals with spinal cord injury. The investigators hypothesize that the blended onsite and telehealth program will achieve better gains in fitness, dietary control, body composition, and pain management scores across a one-year period in comparison to the telehealth-only group. The secondary objective of this study is to examine changes in psychosocial mediators between the two groups to determine if key social cognitive theory constructs were significantly different between the two groups. The investigators hypothesize that the blended onsite and telehealth program will achieve better improvements in these outcomes compared to the telehealth only group.

ELIGIBILITY:
Inclusion Criteria:

* SCI ≥ 1 year post injury
* Able to use arms for exercise
* 18-60 years old
* Reliable access to the internet
* Ability to prepare own food, or have input into person responsible for food preparation
* Can provide own self-care.

Exclusion Criteria:

* Cognitive impairment
* Depression
* Poorly controlled blood pressure (SBP ˃ 159 or DBP ˃ 95 mm HG)
* Cardiovascular disease event within the past six months
* Severe pulmonary disease
* Renal failure
* Current use of insulin or sulfonylurea agents
* Current use of medications for psychosis or bipolar disorder
* Active pressure ulcers

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Change in Warwick-Edinburgh Mental Well-Being Scale Score reflecting resilience | Change from baseline to 7 days post baseline to 1 year post baseline.
  This scale measures resilience-A person's ability to understand, cope, adapt and strive for a positive balance between gains and losses in health and function across their lifespan.

CONTACTS AND LOCATIONS:
Overall Officials: James Rimmer, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Lakeshore Foundation, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided